CLINICAL TRIAL: NCT02717429
Title: Cognitive and Emotion Regulation Training in Multiple Sclerosis
Brief Title: Cognitive and Emotion Regulation Training in MS
Acronym: CERT-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ruchika Prakash, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014H0212
Record Dates: First submitted 2015-10-21; First posted 2016-03-23 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness Meditation Training (MMT) (Experimental): Participants will attend four weekly group mindfulness meditation sessions of a 2-hour duration. The classes are a mixture of experiential practices, discussions surrounding the experiences, and didactics on mindfulness. In addition to the time spent in session, participants will be asked to complete 40 minutes of daily homework, which includes further practice of in-session meditative exercises and brief readings.
  Interventions: Behavioral: Mindfulness Meditation
- Computerized Cognitive Training (Active Comparator): The active control group will be in the form of a cognitive training course where the participants will meet for the same amount of time as the MMT group. Homework will be reading and engaging in cognitive video game exercises for the same duration, around 40 minutes daily, as the MMT group.
  Interventions: Behavioral: Computerized Cognitive Training
- Wait-List Control Group (No Intervention): This group will be used to compare the effects of the two active comparison groups and will not receive any intervention for the four week period.

INTERVENTIONS:
Behavioral: Mindfulness Meditation — The mindfulness meditation-training program is closely modeled after the 8-week mindfulness based stress reduction protocol developed by Dr. Jon Kabat-Zinn. The briefer four weeks of MMT involve the practice of concentrative attention, where different objects are used as the focus of meditative practices. For example, for the first two weeks, the investigators use breath as an anchor for attention. With repeated practices, the objects of sensations, emotions, and thought processes are introduced.
  Arms: Mindfulness Meditation Training (MMT)
Behavioral: Computerized Cognitive Training — The control group, which will be used to compare the effects of mindfulness training on emotional and cognitive functioning of MS patients, will comprise of a cognitive training group, which will provide an attentional-training based approach. In this group, the focus will be to provide the individuals with cognitive training tasks to complete that have been shown to improve attentional ability. The investigators will also discuss relevant MS-related material on cognitive deficits during these courses.
  Arms: Computerized Cognitive Training

SUMMARY:
The investigators propose to conduct a randomized feasibility study of mindfulness meditation training (MMT) relative to an active cognitive training control group and waitlist control group in improving emotional regulation in individuals with MS. Individuals will complete pre- and post-assessments of emotional functioning through a week of daily diary entries, as well as self-report measures and a behavioral paradigm. Additionally, all participants will complete an evaluation of neuropsychological functioning, before and after intervention.

DETAILED DESCRIPTION:
Epidemiological data provides evidence for the manifold increase in rates of depression and anxiety in individuals diagnosed with multiple sclerosis, relative to the general population. Such impaired affective processes, including deficits in emotion regulation have been linked to greater cognitive deficits, a lower quality of life, and greater disease progression in this population. Despite evidence of the deleterious impact of affective functioning on prevalence rates of mood and anxiety disorders; on poor cognitive functioning; and reduced quality of life, much of the targeted intervention research in MS has not directly tested the feasibility, and subsequent efficacy of a psychosocial intervention in improving affective regulation in this population. Thus, the investigators propose to conduct a randomized feasibility study of mindfulness training relative to an active cognitive training control group and waitlist control group in improving emotional regulation in individuals with MS. All individuals that contact the Clinical Neuroscience Laboratory (CNLab) with interest in this study will undergo a phone screening assessing inclusion/exclusion criteria. Those participants meeting I/E criteria will be invited for an online daily diaries portion of the study examining daily engagement in worry and rumination. After completing the week-long daily diary portion of the study, the participant will attend 1-2 in-person pre-assessment sessions, which will also be completed at the completion of the four week intervention. The pre-assessment will involve a thorough assessment of emotion regulation skills, both through self-report questionnaires and behavioral paradigms, and cognitive functioning. Following the assessment sessions, which will be conducted by blind assessors, participants will be randomized to the three groups. The 4-week mindfulness program will be closely modeled after the protocol developed by Dr. Jon Kabat-Zinn, where investigators will have the participants attend once-per-week sessions for 2 hours and complete around 40 minutes a day of homework assignments. The four weeks of mindfulness involve the practice of concentrative attention, where different objects are used as the focus of practices. For example, for the first two weeks, the investigators use breath as an anchor for the mind. With repeated practices, the objects of sensations, emotions, and thought processes are introduced. The classes are a mixture of experiential practices, discussions surrounding the experiences, and didactics on mindfulness. The control group, which will be used to compare the effects of mindfulness training on emotional and cognitive functioning of MS patients, will comprise of a cognitive training group, which will provide an attentional-training based approach. In this group, our focus will be to provide the individuals with cognitive training tasks to complete that have been shown to improve attentional ability. Homework will be reading and practicing using the cognitive video game exercises for the same duration, around 40 minutes daily, as the mindfulness group. Following the four weeks of the intervention, the questionnaires, week-long daily diaries, and behavioral tests from the pretest will be repeated a second time to obtain post-test data for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. 30-59 years of age
2. Score higher than or equal to 23 on the Mini Mental Status Examination (MMSE)
3. Corrected (near and far) visual acuity of 20/40 or better
4. No previous experience with mindfulness or continuous meditation practice
5. Absence of other co-morbid neurological disorders
6. Relapse free for the last 30 days
7. No use of corticosteroids for the last 30 days
8. Clinically definite diagnosis of MS
9. Ability to use a computer and connect the internet from their home
10. Generation of at least two worries and two ruminations during the daily diary portion of the study for the pre-assessment session

Exclusion Criteria:

1. Below 30 years of age or above 59 years of age
2. Score lower than 23 on the MMSE
3. Corrected (near or far) visual acuity of 20/40 or greater
4. Previous experience or participation in a mindfulness program
5. Presence of co-morbid neurological disorders such as:

   * Alzheimers
   * Parkinson's disease
   * Dementia
6. Presence of a relapse within the last 30 days
7. Use of corticosteroids within the last 30 days
8. Clinically isolated syndrome suggestive of MS
9. No ability to use a computer and/or a lack of internet connection from their home
10. No self-generated worries and ruminations in the week-long daily diary portion of the study at pre-assessment

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-10; Primary Completion 2017-05-14 (Actual); Study Completion 2017-05-14 (Actual)

PRIMARY OUTCOMES:
Change in Reported Engagement After Worry and Rumination Inductions | Baseline and 4 weeks
  Participants will engage in worry and rumination inductions during both the pre- and post-intervention sessions. These worries and ruminations will be sampled from the daily diaries participants will fill out 7-days before the pre- and post-intervention sessions. Investigators will be examining the change in emotion and strategy implementation over the course of the worry and rumination inductions. Specifically, investigators will examine the change in reported negative and positive emotion related to the worry and rumination inductions from pre- to post-intervention. Further, investigators will examine the induction-related change in strategy implementation, specifically worry and rumination, over the 4-weeks of intervention.

SECONDARY OUTCOMES:
Cognitive Performance on Brief Repeatable Battery (BRB) | Baseline and 4 weeks
  Participants will perform the entire Brief Repeatable Battery before and after the intervention. Using the categorization developed by Sepulcher (2013), the 5 tests of the BRB will be analyzed using four cognitive domains: attention and executive functioning, verbal memory, visual memory, and word fluency. Based on the computerized cognitive training protocol employed in the current study, investigators hypothesize changes in attention and executive functioning along with visual memory in participants in the cognitive training group, followed by participants in the MMT group compared with the wait-list control participants.
Heart Rate Variability (HRV) | Baseline and 4 weeks
  HRV data will be collected during worry and rumination inductions, as participants regulate their emotions, and at rest.
Daily Emotion Regulation Diary | Baseline and 4 weeks
  Participants will be asked to fill out worry and ruminations using a diary-based methodology a week before the pre-intervention behavioral session and one week after the post-intervention sessions. Changes in average self-reported worry and rumination intensity, emotion regulation strategy use, and successful emotion regulation strategy implementation will be examined as a function of the intervention.
Improvements on a Self-Report Measure of Emotion Dysregulation | Baseline and 4 weeks
  Emotion Dysregulation will be assessed using the Difficulties in Emotion Regulation Scale (DERS). Changes on the total score and sub-facets of DERS will be examined as a function of the intervention.
Improvements on a Self-Report Measure of Depression | Baseline and 4 weeks
  Participants will be administered Beck Depression Inventory before and after the intervention. Change on this measure will be examined to assess the impact of the interventions on symptoms of depression.
Improvements on a Self-Report Measures of Anxiety | Baseline and 4 weeks
  Participants will be administered Penn State Worry Questionnaire before and after the intervention. Change on this measure will be examined to assess the impact of the interventions on symptoms of worry.
Improvements on a Self-Report Measure of Perceived Stress | Baseline and 4 weeks
  Participants will be administered the Perceived Stress Scale before and after the intervention. Changes in these measures will be examined as a function of the intervention.
Improvements on a Self-Report Measure of Quality of Life | Baseline and 4 weeks
  Participants will be administered the Satisfaction with Life Scale before and after the intervention. Change in scores of this measure will be examined to assess changes in quality of life as a function of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika S Prakash, PhD, Principal Investigator — Ohio State University
Locations (1):
- Department of Psychology, The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duraney EJ, Fisher ME, Manglani HR, Andridge RR, Nicholas JA, Prakash RS. Impact of mindfulness training on emotion regulation in multiple sclerosis: Secondary analysis of a pilot randomized controlled trial. Rehabil Psychol. 2022 Nov;67(4):449-460. doi: 10.1037/rep0000456. Epub 2022 Jul 28. PMID 35901401
- [Derived] Schirda B, Duraney E, Lee HK, Manglani HR, Andridge RR, Plate A, Nicholas JA, Prakash RS. Mindfulness training for emotion dysregulation in multiple sclerosis: A pilot randomized controlled trial. Rehabil Psychol. 2020 Aug;65(3):206-218. doi: 10.1037/rep0000324. Epub 2020 May 7. PMID 32378922
- [Derived] Manglani HR, Samimy S, Schirda B, Nicholas JA, Prakash RS. Effects of 4-week mindfulness training versus adaptive cognitive training on processing speed and working memory in multiple sclerosis. Neuropsychology. 2020 Jul;34(5):591-604. doi: 10.1037/neu0000633. Epub 2020 Apr 30. PMID 32352832